CLINICAL TRIAL: NCT06570603
Title: Targeting Components of Distress Tolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jennifer C Veilleux, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R15MH136626-01 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-08-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Distress, Emotional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Psychoeducational Control (Placebo Comparator): Participants will receive psychoeducation only
  Interventions: Behavioral: Psychoeducation
- Self-Efficacy (Only) (Experimental): Single session intervention focusing on increasing self-efficacy to manage distress. Will include brief psychoeducation about emotion, then a focus on agency and self-criticism, using stressors the participant provided from the previous week, with an aim to teach self-compassion skills that will improve self-efficacy.
  Interventions: Behavioral: Self-Efficacy; Behavioral: Psychoeducation
- Willingness (Only) (Experimental): Single session intervention focused on increasing willingness to allow distress. Will include brief psychoeducation about emotion, then a discussion of values and how allowing and experiencing emotions nourishes values, experiencing discomfort enhances growth. Will use stressors from the prior week as examples.
  Interventions: Behavioral: Willingness; Behavioral: Psychoeducation
- Combined Willingness and Self-Efficacy (Experimental): Single session intervention focused on increasing both willingness and self-efficacy. Will include brief psychoeducation about emotion, then a combination of using values and self-compassion to increase both allowing and self-efficacy.
  Interventions: Behavioral: Self-Efficacy; Behavioral: Willingness; Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Self-Efficacy — Brief skills based psychotherapy session to increase perceived self-efficacy for withstanding distress, giving participants increased beliefs that they *can* do it.
  Arms: Combined Willingness and Self-Efficacy; Self-Efficacy (Only)
Behavioral: Willingness — Brief skills based psychotherapy session to increase perceived willingness to engage with distress for withstanding distress, giving participants increased motivation to try.
  Arms: Combined Willingness and Self-Efficacy; Willingness (Only)
Behavioral: Psychoeducation — Psychoeducation about the components and functions of emotion.

SUMMARY:
The goal of this clinical trial is to learn which aspects of distress intolerance (i.e., difficulties withstanding upsetting emotional states) are the most important for improving effective emotion regulation and associated mental health symptoms.

The main questions it aims to answer are:

How are willingness to feel upset and self-efficacy for withstanding distress associated with different emotion regulation strategies used in daily life?

Does targeting willingness to feel upset and/or self-efficacy for withstanding distress help people use more effective emotion regulation strategies in daily life when they feel upset?

Are improvements in emotion regulation strategies in daily life associated with fewer symptoms of mental health problems over time?

Participants will:

Answer questions about their moods, willingness to feel upset, self-efficacy for withstanding distress and emotion regulation strategies for three weeks using a cell phone app

Undergo a willingness, self-efficacy, combined or psychoeducational control intervention in the lab

Be prompted to use the intervention skill via the cell phone app during the second week, after the intervention

Complete weekly reports of mental health symptoms

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Uses Android or iPhone smartphone
* Depression Anxiety and Stress Scale (DASS-21) scores of 42 and higher
* Distress Intolerance Index (DII) scores of 3 or higher

Exclusion Criteria:

* Work or School that does not allow consistent access to phone (or is unsafe)
* No internet access for completing follow-up surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Engagement behaviors | Assessed 5x/day via ecological momentary assessment
  Emotion regulation strategies reflective of engagement; these are new items developed for this study and are not from an established scale. All items will be rated from 0 (not at all) to 6 (extremely). There will be 7 items assessing labeling ("I'm using emotion words to describe how I feel right now"), processing ("I'm reflecting on or writing about my feelings"), sharing ("I'm sharing how I feel with another person"), physical feeling ("I'm intentionally feeling my feelings in my body"), curiously considering ("I'm curiously considering how my feelings came about"), defusion ("I'm observing my feelings without getting 'stuck' in them"), and importance ("I'm trying to think about how this current situation maps on to what matters.")
Disengagement behaviors | Assessed 5x/day via ecological momentary assessment
  Emotion regulation strategies reflective of disengagement, some of which were modified from a momentary experiential avoidance measure (Hershenberg et al., 2017). All items will be rated from 0 (not at all) to 6 (extremely).Items will assess distraction ("Trying to distract myself from my feelings'), thought suppression ("Trying to push unwanted thoughts out of my mind."), discounting ("I'm telling myself I shouldn't be feeling the way I'm feeling"), expressive suppression ("I'm trying to control my feelings by not expressing them"), procrastination ("I'm intentionally putting of an unpleasant task until later"), denial ("I'm trying to 'turn off' the feelings that I don't want to feel"), and reduce importance ("Trying to think about the current situation as unimportant to me.")
GAD-7 | Baseline, weekly for three weeks and then after one month followup
  Symptoms of anxiety
PHQ-9 | Baseline, weekly for three weeks and then after one month followup
  symptoms of depression
AUDIT | Baseline, weekly for three weeks and then after one month followup
  Alcohol misuse
Binge Eating Disorder Scale | Baseline, weekly for three weeks and then after one month followup
  binge eating symptoms
DSM Cross-Cutting Symptom Measure | Baseline, weekly for three weeks and then after one month followup
  symptoms of psychopathology

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS) | Baseline, weekly for three weeks and then after one month followup
  life satisfaction
Self-Compassion Scale - Short | Baseline, weekly for three weeks and then after one month followup
  self-criticism and self-compassion
State Loss of Interest and Pleasure Scale | Baseline, weekly for three weeks and then after one month followup
  anhedonia
Rumination and Reflection Questionnaire | Baseline, weekly for three weeks and then after one month followup
  rumination and self-reflective tendencies

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas - Fayetteville, Fayetteville, Arkansas, United States